CLINICAL TRIAL: NCT00499746
Title: Medications Development for Drug Abuse Disorders
Brief Title: The Discriminative Effects of Tramadol in Humans
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Eric Strain, MD, Professor, Johns Hopkins University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NIDA-18125-3; R01DA018125 (NIH); DPMCDA (Other: NIDA)
Record Dates: First submitted 2007-07-09; First posted 2007-07-11 (Estimated); Results first posted 2017-10-17 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2017-09

CONDITIONS: Opioid Abuse; Opioid Addiction; Stimulant Abuse; Stimulant Addiction
Keywords: drug discrimination; opioid pharmacology; behavioral pharmacology; human research
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Tramadol; Sugars; Hydromorphone; Methylphenidate; Central Nervous System Stimulants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Tramadol (Active Comparator): oral dose, once per day
  Interventions: Drug: tramadol
- Placebo (Placebo Comparator): oral dose, once per day
  Interventions: Drug: placebo
- hydromorphone (Active Comparator): oral dose, once per day
  Interventions: Drug: Hydromorphone
- methylphenidate (Active Comparator): oral dose, once per day
  Interventions: Drug: Methylphenidate

INTERVENTIONS:
Drug: tramadol — oral dose, once per day
  Other Names: Ultram
  Arms: Tramadol
Drug: placebo — oral dose, once per day
  Other Names: sugar pill
  Arms: Placebo
Drug: Hydromorphone — oral dose, once per day
  Other Names: Dilaudid
  Arms: hydromorphone
Drug: Methylphenidate — oral dose, once per day
  Other Names: stimulant
  Arms: methylphenidate

SUMMARY:
This research is part of a set of studies whose purpose is to test whether tramadol can be used for the treatment of opioid addiction. Tramadol is already available in the United States as a pain medicine marketed as Ultram. It has effects similar to morphine, and it may also have effects similar to other drugs like stimulants. The doses of tramadol used in this study are higher than those generally used for the treatment of pain. To be in this study a participant must be a user of opioids (drugs like heroin) and stimulants (drugs like cocaine), but cannot be addicted to either. The person must be between 21-55 years old, and generally healthy. Up to 12 people will take part in this study.

DETAILED DESCRIPTION:
This is a human laboratory study that tests the effects of tramadol as a step in the possible development of this medication as a new treatment for opioid dependence. Tramadol is a mild/moderate mu agonist opioid currently marketed as an analgesic that has a unique profile of effects. One of the primary metabolites of tramadol, mono-O-demethyltramadol (referred to as M1) exerts opioid agonist effects at the mu receptor. In addition, tramadol and M1 produce reuptake blockade of monoamines, and this latter effect may positively influence its analgesic efficacy, in addition to influencing the subjective effects produced by tramadol. Preclinical evidence suggests that tramadol's effects on monoamine reuptake may have antidepressant qualities as well. Given tramadol's diverse pharmacodynamic profile, a systematic characterization of its subjective effects in opioid-experienced subjects would provide valuable information regarding its abuse liability, and its potential utility as a treatment for opioid dependence.

The characterization of an opioid medication's profile can be accomplished through a variety of experimental procedures. One useful procedure for assessing the profile of an opioid is a drug discrimination procedure. In this methodology, subjects are first trained to discriminate reference drugs such as placebo and an opioid agonist, and then administered doses of a novel compound to determine how like (or unlike) it is to the reference training conditions. Our laboratory has a long history of using this drug discrimination methodology to study and to characterize opioids with varying opioid receptor activity profiles. Studies have generally included either two or three training conditions in humans. Using this technique in volunteers, studies have characterized the profile of a number of opioids including (for example) butorphanol, nalbuphine, pentazocine, and buprenorphine.

While most of these studies testing the effects of mixed agonist-antagonist opioids have used an opioid agonist and placebo as the training conditions, tramadol's profile of effects suggests that there may be a non-opioid component of action at serotonin and norepinephrine sites that will be useful to distinguish. In particular, it is of interest to determine the extent to which tramadol is identified as being like a prototypic mu agonist opioid, whether it is substantially identified as being like a non-opioid compound, and if this non-opioid component is related to enhancement of monoamine effects. In order to provide a meaningful non-opioid contrast training condition, this study will compare different doses of tramadol to training conditions of placebo, a mu agonist opioid, and a prototypic stimulant.

Overall, this evaluation will provide a greater understanding of the subjective effect profile of tramadol in comparison to a prototypic mu opioid and a prototypic stimulant. If tramadol is to be useful in the treatment of opioid dependence, a thorough assessment of its subjective effects in experienced opioid and stimulant abusers is warranted.

ELIGIBILITY:
Inclusion Criteria:

* Study subjects are male and female non-dependent opioid users with active stimulant use.
* Between the ages of 21-55
* In good physical health
* Without significant psychiatric illness besides their drug use.
* Females are required to provide a negative pregnancy test prior to study participation.

Exclusion Criteria:

* Subjects are excluded if they have evidence of significant medical (e.g., insulin dependent diabetes mellitus) or psychiatric (e.g., schizophrenia) illness.
* Subjects with a history of seizures will be excluded.
* Persons with current history of significant alcohol or sedative/hypnotic drug use will be excluded from study participation.
* Applicants seeking treatment for their substance abuse will not be admitted to the study, and will be provided information about treatment services available.

Ages: 21 Months to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2007-11; Primary Completion 2010-04 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric C Strain, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States

REFERENCES:
- [Result] Duke AN, Bigelow GE, Lanier RK, Strain EC. Discriminative stimulus effects of tramadol in humans. J Pharmacol Exp Ther. 2011 Jul;338(1):255-62. doi: 10.1124/jpet.111.181131. Epub 2011 Apr 5. PMID 21467190

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Participant flow is reported in single group due to the number of randomized sequences. In Phase 1 and Phase 2, each participant received two exposures of each training drug in randomize order (placebo, Hydromorphone 8 mg, Methylphenidate 60 mg). In Phase 3, each participant received randomized exposure to placebo, Hydromorphone (4 and 8 mg), Methylphenidate (30 and 60 mg), tramadol (50, 100, 200, and 400 mg).
Period: Phase 1(6-9 One Day Sessions)
Arm/Group | All Participants
Started | 20
Completed | 8
Not Completed | 12
Not completed — Failed to perform study task | 7
Not completed — Withdrawal by Subject | 3
Not completed — Investigator decision | 1
Not completed — Unable to determine | 1
Period: Phase 2 (6-9 One Day Sessions)
Arm/Group | All Participants
Started | 8
Completed | 8
Not Completed | 0
Period: Phase 3 (9-14 One Day Sessions)
Arm/Group | All Participants
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Acquisition of Discrimination Assessed by Accuracy of the Discrimination Test
Description: The acquisition of discrimination was to test whether volunteers could identify each training drug condition by the correct letter code. Results are the percentage of correct responses with a range of 0% to 100%.
Time Frame: 1 day
Measure: Mean (Full Range); unit: percent of correct response
Arm/Group | Placebo 0 mg | Hydromorphone 8 mg | Methylphenidate 60 mg
Number analyzed (Participants) | 8 | 8 | 8
percent of correct response | 87 [0 to 100] | 87.5 [0 to 100] | 90 [0 to 100]

2. Primary Outcome: Discrimination Effects Assessed by Operant Responses
Description: Volunteers emitted operant responses on computer keys that corresponded to the training letter, on a fixed interval 1 second schedule for 8.5 minutes. The range is from 0 to 500 operant responses.
Time Frame: 1 day
Measure: Mean (Standard Error); unit: Responses
Arm/Group | Placebo 0 mg | Hydromorphone 4 mg | Hydromorphone 8 mg | Methylphenidate 30 mg | Methylphenidate 60 mg | Tramadol 50 mg | Tramadol 100 mg | Tramadol 200 mg | Tramadol 400 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
Responses
  Placebo | 455.5 (9.6) | 116.6 (76.4) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 464.1 (4.2) | 341.3 (74.8) | 86.6 (62.0) | 115.6 (75.7)
  Hydromorphone | 0.0 (0.0) | 341.3 (74.7) | 453.4 (9.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 118.1 (77.3) | 367.0 (60.2) | 282.9 (83.4)
  Methylphenidate | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 465.4 (4.7) | 465.8 (3.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 59.9 (59.9)

3. Primary Outcome: Discrimination Effects Assessed by Point Distribution
Description: In point distribution, volunteers distributed 50 points among three training drug letters depending on how certain they were of the identity of the administrated drug. Maximum total is 50 points.
Time Frame: 1day
Measure: Mean (Standard Error); unit: Points distributed
Arm/Group | Placebo 0 mg | Hydromorphone 4 mg | Hydromorphone 8 mg | Methylphenidate 30 mg | Methylphenidate 60 mg | Tramadol 50 mg | Tramadol 100 mg | Tramadol 200 mg | Tramadol 400 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
Points distributed
  Placebo | 50.0 (0.0) | 11.9 (7.8) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 50.0 (0.0) | 37.5 (8.2) | 9.4 (6.6) | 12.5 (8.2)
  Hydromorphone | 0.0 (0.0) | 38.1 (7.8) | 50.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 12.5 (8.2) | 38.3 (6.5) | 31.3 (9.1)
  Methylphenidate | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 50.0 (0.0) | 50.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 6.3 (6.3)

4. Primary Outcome: Discrimination Effects Assessed by Discrete Choice
Description: During discrete choice, volunteers were given three choices (placebo, hydromorphone, methylphenidate) and were asked to choose which of the training drugs they thought they received. The outcome measure illustrates the percentage of participants who chose either placebo, hydromorphone, or methylphenidate during each drug condition (i.e., Placebo, Hydromorphone 8 mg, Tramadol 50 mg, etc.), ranging from 0-100.
  The outcome measure represents the percentage of participants who chose either placebo, opioid agonist, or stimulant across each drug condition.
Time Frame: 1 day
Measure: Number; unit: percentage of drug identification
Arm/Group | Placebo 0 mg | Hydromorphone 4 mg | Hydromorphone 8 mg | Methylphenidate 30 mg | Methylphenidate 60 mg | Tramadol 50 mg | Tramadol 100 mg | Tramadol 200 mg | Tramadol 400 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
percentage of drug identification
  Placebo | 100 | 25 | 0 | 0 | 0 | 100 | 75 | 25 | 25
  Hydromorphone | 0 | 75 | 100 | 0 | 0 | 0 | 25 | 75 | 63
  Methylphenidate | 0 | 0 | 0 | 100 | 100 | 0 | 0 | 0 | 12

5. Secondary Outcome: Physiologic Effects Assessed by the Pharmacological Class Questionnaire
Description: During the peak (assessed at 120 min) of each drug administration, participants were asked to complete the pharmacological class questionnaire. The pharmacological class questionnaire had volunteers indicate which drug class was most similar to the drug condition they received. Ten drug classes were listed with descriptive labels and examples of each: placebo, opiates (or opioid agonist), phenothiazines, barbiturates, antidepressants, opiate antagonists, hallucinogens, benzodiazepines, stimulants, and other. Of these choices, participants chose 3: placebo, opioid agonist, and stimulant.
  The outcome measure represents the percentage of participants who chose either placebo, opioid agonist, or stimulant across each drug condition.
Time Frame: Measure at 120 min after drug administration
Measure: Number; unit: percentage of drug identification
Arm/Group | Placebo 0 mg | Hydromorphone 4 mg | Hydromorphone 8 mg | Methylphenidate 30 mg | Methylphenidate 60 mg | Tramadol 50 mg | Tramadol 100 mg | Tramadol 200 mg | Tramadol 400 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
percentage of drug identification
  Placebo | 100 | 25 | 0 | 0 | 0 | 100 | 75 | 37 | 25
  Opioid Agonist | 0 | 75 | 100 | 0 | 0 | 0 | 25 | 63 | 63
  Stimulant | 0 | 0 | 0 | 100 | 100 | 0 | 0 | 0 | 12

6. Secondary Outcome: Physiological Effects Assessed by Peak Change From Baseline Pupil Diameter
Description: Change in pupil diameter (mm) at peak (120 min) compared to baseline measure of pupil diameter
Time Frame: Measure at 120 min after drug administration
Measure: Mean (Standard Error); unit: mm
Arm/Group | Placebo 0 mg | Hydromorphone 4 mg | Hydromorphone 8 mg | Methylphenidate 30 mg | Methylphenidate 60 mg | Tramadol 50 mg | Tramadol 100 mg | Tramadol 200 mg | Tramadol 400 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
mm | -0.5 (0.2) | -1.2 (0.2) | -1.9 (0.2) | -0.6 (0.3) | -0.3 (0.2) | -0.5 (0.1) | -0.2 (0.1) | -0.8 (0.3) | -0.8 (0.3)

7. Secondary Outcome: Peak Change From Baseline Opioid Agonist Effects Assessed by the Visual Analog Scale (VAS)
Description: The Visual Analog Scale (VAS) measures subjective ratings of opioid agonist effects. The scale on this measure ranges from 0 being "Not at all" to 100 being "Extremely". On this scale, higher scores indicate a stronger drug effect. The outcome measure illustrates a difference from peak (120 min) to baseline measure on VAS.
Time Frame: Measure at 120 min after drug administration
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo 0 mg | Hydromorphone 4 mg | Hydromorphone 8 mg | Methylphenidate 30 mg | Methylphenidate 60 mg | Tramadol 50 mg | Tramadol 100 mg | Tramadol 200 mg | Tramadol 400 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
units on a scale | 1.4 (0.7) | 2.9 (1.0) | 4.8 (2.1) | 2.1 (0.5) | 3.4 (1.2) | 0.4 (0.4) | 1.6 (0.7) | 2.1 (1.0) | 3.8 (1.8)

8. Secondary Outcome: Peak Change From Baseline Stimulant Effects Assessed by the Visual Analog Scale (VAS)
Description: The Visual Analog Scale (VAS) measures subjective ratings of stimulant effects. The scale on this measure ranges from 0 being "Not at all" to 100 being "Extremely". On this scale, higher scores indicate a stronger drug effect. The outcome measure illustrates a difference from peak (120 min) to baseline measure.
Time Frame: Measure at 120 min after drug administration
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo 0 mg | Hydromorphone 4 mg | Hydromorphone 8 mg | Methylphenidate 30 mg | Methylphenidate 60 mg | Tramadol 50 mg | Tramadol 100 mg | Tramadol 200 mg | Tramadol 400 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
units on a scale | 1.4 (0.8) | 3.6 (1.0) | 3.6 (1.2) | 8.0 (1.6) | 10.6 (2.3) | 0.6 (0.4) | 0.9 (0.5) | 4.9 (2.0) | 6.9 (2.1)

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No